CLINICAL TRIAL: NCT02845921
Title: Comparison of Leg Elevation and Leg Wrapping in the Prevention of Propofol Induced Hypotension: A Prospective Randomised Controlled Study
Brief Title: Comparison of Leg Elevation and Leg Wrapping in the Prevention of Propofol Induced Hypotension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nitte University (Other)
Responsible Party: Principal Investigator, Dr. Sara Jaison, Junior Resident, Nitte University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INST.EC/EC/066/2015-16
Record Dates: First submitted 2016-06-30; First posted 2016-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Propofol Induced Hypotension
Keywords: Propofol; Hypotension; Induction of anaesthesia; Leg elevation; Leg wrapping
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group C Control (Placebo Comparator): Patient will be shifted to operation theatre. Electrocardiography (ECG), pulse oximeter and non-invasive blood pressure (NIBP) monitors will be attached. Baseline vitals will be noted. Intravenous access will be secured and crystalloids at 100ml/hr will be given. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be neither elevated or wrapped. Vitals will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Muscle relaxation will be achieved by inj. vecuronium 0.1mg/kg body weight. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube.
  Interventions: Other: control
- Group E Leg elevation (Experimental): Patient will be shifted to operation theatre. Crystalloids at 100ml/hr will be given. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs are elevated and supported on a stand making an angle of 30 degree to the horizontal. Vitals will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Muscle relaxation will be achieved by inj. vecuronium 0.1mg/kg body weight. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Stand will be removed and legs will be brought to horizontal position 10 minutes after intubation.
  Interventions: Other: leg elevation
- Group W Leg wrapping (Experimental): Patient will be shifted to operation theatre. Crystalloids at 100ml/hr will be given. Analgesia will be given by inj fentanyl. Each lower limb will be elevated alternately and wrapped from toe to mid-thigh with Esmarch bandage. Care will be taken to avoid compressing the legs to greater than arterial pressure by confirming the presence of pulse using a saturation probe. Following wrapping, the lower limbs will be brought to horizontal position. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol injected over 30 seconds. Muscle relaxation by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Esmarch bandage will be removed 10 minutes after intubation.
  Interventions: Other: leg wrapping

INTERVENTIONS:
Other: leg elevation — A stand making an angle of 30 degree to the horizontal is used to elevate both the legs
  Arms: Group E Leg elevation
Other: leg wrapping — Esmarch bandage is used to wrap each lower limb
  Arms: Group W Leg wrapping
Other: control — no intervention has been done
  Arms: Group C Control

SUMMARY:
Propofol is an intravenous anaesthetic agent used for both induction and maintenance of anaesthesia. An important adverse effect is the significant fall in blood pressure. The current clinical study will be done to determine the efficacy of leg elevation and wrapping in reducing the incidence and severity of propofol induced hypotension in patients undergoing general anaesthesia.

DETAILED DESCRIPTION:
Propofol is an intravenous anaesthetic agent used for both induction and maintenance of anaesthesia. It is widely employed due to its quick onset of action, short half life and rapid recovery. An important adverse effect is the significant fall in blood pressure. Although the exact mechanism of propofol induced hypotension is not known, venodilation, decreased peripheral resistance and decrease in cardiac output has been suggested.2 Though the hypotension is transient, it can produce devastating effects. Hence there is a need to prevent it. Moreover, several attempts at treating propofol induced hypotension have been met with variable and limited success.

Hypotension following spinal anaesthesia is also a frequent problem. It is generally treated with intravenous fluids and vasopressors. Simple and non pharmacological measures like leg elevation and leg wrapping with Esmarch bandage were reported to be successful.3 These reduce the incidence and severity of hypotension associated with spinal anaesthesia by improving the venous return.

The mechanisms of hypotension following intravenous propofol and spinal anaesthesia are almost similar. Therefore, the investigators hypothesize that leg elevation and wrapping can be attempted to reduce propofol induced hypotension. They are simple and cost effective techniques that will reduce the need for pharmacological measures to control hypotension. As the literature search did not reveal any information regarding the usefulness of these techniques in propofol induced hypotension, the current clinical study will be done to determine the efficacy of leg elevation and wrapping in reducing the incidence and severity of propofol induced hypotension in patients undergoing general anaesthesia.

The current study will compare the efficacy of leg elevation and leg wrapping in reducing the incidence and severity of propofol induced hypotension in terms of incidence of hypotension, magnitude of decrease in systolic, diastolic and mean arterial blood pressures, need for pharmacological measures to treat hypotension, changes in heart rate and adverse clinical outcomes, if any. It will be a prospective randomised controlled open label study from January 2016 to August 2017 involving 150 adult patients undergoing general anaesthesia.

For statistical analysis, descriptive statistics - minimum, maximum, mean and standard deviation will be used. Independent sample t test for data following normal distribution and for data not following normal distribution, Mann-Whitney U test will be used. P value less than 0.05 will be considered statistically significant. To study relationship between hypotension and other variables, Pearson's correlation will be used. Confidence interval will be calculated to 95%.

ELIGIBILITY:
Inclusion Criteria:

* Patients belonging to ASA physical status I and II undergoing endotracheal general anaesthesia

Exclusion Criteria:

* Patient refusal
* Contraindication to application of bandage
* Partial or complete limb amputation
* Difficult airway
* Use of extraglottic airway device
* Pregnancy
* On antihypertensive or vasoactive medication
* Autonomic neuropathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
incidence of hypotension at baseline | baseline
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 0 minutes after leg elevation or wrapping | 0 minutes after leg elevation or wrapping
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 0 minutes after induction with propofol | 0 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 1 minute after induction | 1 minute after induction
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 2 minutes after induction | 2 minutes after induction
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 3 minutes after induction | 3 minutes after induction
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 4 minutes after induction | 4 minutes after induction
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 5 minutes after induction | 5 minutes after induction
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 0 minutes after intubation | 0 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 1 minute after intubation | 1 minute after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 2 minutes after intubation | 2 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 3 minutes after intubation | 3 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 4 minutes after intubation | 4 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 5 minutes after intubation | 5 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 6 minutes after intubation | 6 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 7 minutes after intubation | 7 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 8 minutes after intubation | 8 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 9 minutes after intubation | 9 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.
incidence of hypotension at 10 minutes after intubation | 10 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline blood pressure including systolic, diastolic and mean arterial blood pressures will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Blood pressures will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Blood pressures will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Hypotension will be defined as a drop in systolic blood pressure to less than 30% of baseline values or to MAP <60mm Hg. Incidence of hypotension will be noted.

SECONDARY OUTCOMES:
Magnitude of change in systolic blood pressure from baseline at 0 minutes after leg leg elevation or wrapping | baseline, after leg elevation or wrapping
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 0 minutes after induction | baseline, at 0 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 1 minute after induction | baseline, at 1 minute after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 2 minutes after induction | baseline, at 2 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 3 minutes after induction | baseline, at 3 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 4 minutes after induction | baseline, at 4 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 5 minutes after induction | baseline, at 5 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 0 minutes after intubation | baseline, at 0 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 1 minute after intubation | baseline, at 1 minute after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 2 minutes after intubation | baseline, at 2 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 3 minutes after intubation | baseline, at 3 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 4 minutes after intubation | baseline, at 4 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 5 minutes after intubation | baseline, at 5 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 6 minutes after intubation | baseline, at 6 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 7 minutes after intubation | baseline, at 7 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 8 minutes after intubation | baseline, at 8 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 9 minutes after intubation | baseline, at 9 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in systolic blood pressure from baseline at 10 minutes after intubation | baseline, at 10 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline systolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Systolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Systolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Systolic blood pressure will be recorded every minute till 10 min post intubation. Magnitude of change in systolic blood pressure from baseline will be noted
Magnitude of change in diastolic blood pressure from baseline at 0 minutes after leg elevation or wrapping | baseline, at 0 minutes after leg elevation or wrapping, at induction with propofol, every minute till 5 minutes after induction, at intubation and every minute thereafter upto 10 min post intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 0 minutes after induction with propofol | baseline, at 0 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 1 minute after induction with propofol | baseline, at 1 minute after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 2 minutes after induction with propofol | baseline, at 2 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 3 minutes after induction with propofol | baseline, at 3 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 4 minutes after induction with propofol | baseline, at 4 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 5 minutes after induction with propofol | baseline, at 5 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 0 minutes after intubation | baseline, at 0 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 1 minute after intubation | baseline, at 1 minute after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 2 minutes after intubation | baseline, at 2 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 3 minutes after intubation | baseline, at 3 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 4 minutes after intubation | baseline, at 4 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 5 minutes after intubation | baseline, at 5 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 6 minutes after intubation | baseline, at 6 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 7 minutes after intubation | baseline, at 7 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 8 minutes after intubation | baseline, at 8 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 9 minutes after intubation | baseline, at 9 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in diastolic blood pressure from baseline at 10 minutes after intubation | baseline, at 10 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline diastolic blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Diastolic blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Diastolic blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in diastolic blood pressure from baseline will be noted.
Magnitude of change in mean arterial blood pressure from baseline at 0 minutes after leg elevation or wrapping | baseline, 0 minutes after leg elevation or wrapping
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 1 minute after induction with propofol | baseline, 0 minute after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 2 minutes after induction with propofol | baseline, 2 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 3 minutes after induction with propofol | baseline, 3 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 4 minutes after induction with propofol | baseline, 4 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 5 minutes after induction with propofol | baseline, 5 minutes after induction with propofol
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 0 minute after intubation | baseline, 0 minute after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 1 minutes after intubation | baseline, 1 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 2 minutes after intubation | baseline, 2 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 3 minutes after intubation | baseline, 3 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 4 minutes after intubation | baseline, 4 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 5 minutes after intubation | baseline, 5 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 6 minutes after intubation | baseline, 6 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 7 minutes after intubation | baseline, 7 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 8 minutes after intubation | baseline, 8 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 9 minutes after intubation | baseline, 9 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
Magnitude of change in mean arterial blood pressure from baseline at 10 minutes after intubation | baseline, 10 minutes after intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. Mean arterial blood pressure will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Mean arterial blood pressure will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Magnitude of change in mean arterial blood pressure from baseline will be noted
changes in heart rate from baseline at 0 minutes after leg elevation or wrapping | baseline, 0 minutes after leg elevation or wrapping
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 0 minutes after induction with propofol | baseline, 0 minute after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 1 minutes after induction with propofol | baseline, 1 minutes after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 2 minutes after induction with propofol | baseline, 2 minutes after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 3 minutes after induction with propofol | baseline, 3 minutes after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 4 minutes after induction with propofol | baseline, 4 minutes after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 5 minutes after induction with propofol | baseline, 5 minutes after induction with propofol
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 0 minutes after intubation | baseline, 0 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 1 minute after intubation | baseline, 1 minute after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 2 minutes after intubation | baseline, 2 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 3 minutes after intubation | baseline, 3 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 4 minutes after intubation | baseline, 4 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 5 minutes after intubation | baseline, 5 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 6 minutes after intubation | baseline, 6 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 7 minutes after intubation | baseline, 7 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 8 minutes after intubation | baseline, 8 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 9 minutes after intubation | baseline, 9 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted
changes in heart rate from baseline at 10 minutes after intubation | baseline, 10 minutes after intubation
  Patient will be shifted to operation theatre. Baseline heart rate will be noted. Analgesia will be given by inj fentanyl 2µg/kg body weight. Lower limbs will be elevated, wrapped or none according to group allocation. Heart rate will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol 2mg/kg body weight injected over 30 seconds. Heart rate will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation will be achieved by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed with appropriate sized endotracheal tube. Heart rate will be recorded every minute till 10 min post intubation. Changes in heart rate from baseline will be noted

OTHER OUTCOMES:
Need for pharmacological measures to treat hypotension | baseline, after leg elevation or wrapping, at induction with propofol, every minute till 5 minutes after induction, at intubation and every minute thereafter upto 10 min post intubation
  Patient will be shifted to operation theatre. Non-invasive blood pressure (NIBP) monitor will be attached. Baseline mean arterial blood pressure (MAP) will be noted. Analgesia will be given by inj fentanyl. Lower limbs will be elevated, wrapped or none according to group allocation. MAP will be recorded again. 3 minutes of pre-oxygenation will be done. Anaesthesia will be induced with inj. propofol. MAP will be noted at induction with propofol and for every minute till 5 minutes after induction. Muscle relaxation by inj. vecuronium. Patient will be ventilated with oxygen for 5 minutes. Orotracheal intubation will be performed. MAP<55mm Hg will be treated by rapid intravenous fluid administration and by intravenous mephentermine 6mg bolus increments every minute until the systolic pressure rises to greater than 70% of baseline or to above 90mm Hg. Total dose of mephentermine required will be noted.
Tachycardia | baseline, after leg elevation or wrapping, at induction with propofol, every minute till 5 minutes after induction, at intubation and every minute thereafter upto 10 min post intubation
  Tachycardia will be defined as heart rate more than 100bpm or increase by more than 30% over baseline value. Any incidence of tachycardia during the procedure will be noted
Bradycardia | baseline, after leg elevation or wrapping, at induction with propofol, every minute till 5 minutes after induction, at intubation and every minute thereafter upto 10 min post intubation
  Bradycardia will be defined as heart rate less than 50bpm or decrease by more than 30% below baseline value. Any incidence of bradycardia during the procedure will be noted
Arrhythmia | baseline, after leg elevation or wrapping, at induction with propofol, every minute till 5 minutes after induction, at intubation and every minute thereafter upto 10 min post intubation
  any incidence of arrhythmia during the procedure will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Sripada G Mehandale, MBBS, MD, Study Director — Associate Professor
Locations (1):
- Justice K. S. Hegde Hospital, K S Hegde Medical Academy, Nitte University, Mangalore, Dakshina Kannada, India

IPD SHARING:
Plan to Share IPD: Yes
Age, sex, weight, diagnosis, surgery, asa physical status, heart rate, systolic blood pressure, diastolic blood pressure, mean arterial pressure

REFERENCES:
- [Background] McNeir DA, Mainous EG, Trieger N. Propofol as an intravenous agent in general anesthesia and conscious sedation. Anesth Prog. 1988 Jul-Aug;35(4):147-51. PMID 3046442
- [Background] Muzi M, Berens RA, Kampine JP, Ebert TJ. Venodilation contributes to propofol-mediated hypotension in humans. Anesth Analg. 1992 Jun;74(6):877-83. doi: 10.1213/00000539-199206000-00017. PMID 1595920
- [Background] Rout CC, Rocke DA, Gouws E. Leg elevation and wrapping in the prevention of hypotension following spinal anaesthesia for elective caesarean section. Anaesthesia. 1993 Apr;48(4):304-8. doi: 10.1111/j.1365-2044.1993.tb06948.x. PMID 8494130
- [Background] Masoudifar M, Beheshtian E. Comparison of cardiovascular response to laryngoscopy and tracheal intubation after induction of anesthesia by Propofol and Etomidate. J Res Med Sci. 2013 Oct;18(10):870-4. PMID 24497858
- [Background] Moller Petrun A, Kamenik M. Bispectral index-guided induction of general anaesthesia in patients undergoing major abdominal surgery using propofol or etomidate: a double-blind, randomized, clinical trial. Br J Anaesth. 2013 Mar;110(3):388-96. doi: 10.1093/bja/aes416. Epub 2012 Nov 19. PMID 23166149
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] Singh K, Payal YS, Sharma JP, Nautiyal R. Evaluation of hemodynamic changes after leg wrapping in elective cesarean section under spinal anesthesia. J Obstet Anaesth Crit Care. 2014;4:23-8